CLINICAL TRIAL: NCT05085704
Title: Brain Metabolism Observed at 7 Tesla in Health and Metabolic Disease.
Brief Title: Brain Metabolism Observed at 7 Tesla
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Juan Pascual, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0560
Record Dates: First submitted 2021-08-31; First posted 2021-10-20 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Glut1 Deficiency Syndrome 1; Glucose Metabolism Disorders; Epilepsy; Glut1 Deficiency Syndrome 1, Autosomal Recessive; Glucose Transporter Type 1 Deficiency Syndrome; Glucose Transporter Protein Type 1 Deficiency Syndrome; Glucose Transport Defect
MeSH Terms: conditions — Glucose Metabolism Disorders; Epilepsy; Glut1 Deficiency Syndrome; Glycogen Storage Disease Id | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Adolescents and adults with Glut1 deficiency: 1. Adolescents and adults with previously documented diagnosis of Glut1 Deficiency with diagnosis genetically confirmed or confirmed by PET scan of the brain.
  2. Ages 16 to 65
  3. Persons with dental fillings, dental crowns, and short (max.4 cm) dental retainer wires can be included.
  Interventions: Device: Magnetic resonance imaging
- Normal healthy adolescents and adults: 1. Adolescents or adults in good general health.
  2. Ages 16 to 65.
  3. Persons with dental fillings, dental crowns, and short (max. 4 cm) dental retainer wires can be included.
  Interventions: Device: Magnetic resonance imaging

INTERVENTIONS:
Device: Magnetic resonance imaging — Medical imaging technique used in radiology to form pictures of the anatomy.
  Other Names: MRI

SUMMARY:
The goal is to develop methodology to monitor flux in the citric acid cycle in brain via 13C nuclear magnetic resonance (NMR) spectroscopy at 7 Tesla.

DETAILED DESCRIPTION:
The goal is to establish a protocol to 13C-label (from 13C-glucose) several physiological molecules: glucose, lactate, pyruvate and derived compounds. All of these molecules can undergo oxidation in the citric acid cycle. The intent is to study the 13C labeling pattern of these molecules in control and G1D subjects to determine if downstream products (such as 13C bicarbonate or 13C glutamate) due to oxidation in the mitochondria can be detected in brain or in blood by NMR analysis. While inside the instrument, the subjects may also undergo a 7T MR exam to correlate spectroscopy with brain structure.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents and adults with previously documented diagnosis of Glut1 Deficiency with diagnosis genetically confirmed or confirmed by PET scan of the brain.
2. Ages 16 to 65
3. Persons with dental fillings, dental crowns, and short (max.4 cm) dental retainer wires can be included.

Exclusion Criteria:

1. People or patients with uncontrolled seizure disorder, defined as grand mal (not absence) seizure in the preceding 3 months.
2. Pregnant females will be excluded. A serum or urine pregnancy test will be administered to all females of child bearing potential within 24 hours of administration of the tracer and MRI scan. The pregnancy test will be communicated in person by the study PI. Positive results in subjects 17 years old or younger will be disclosed to parent/guardian only.
3. Subjects with typical implanted orthopedic metal in bone may be considered for inclusion in a 7T scan providing the implant is not within the volume of the radio frequency coil. The PI and the AIRC Medical Director will discuss each case and determine eligibility.
4. Persons with ICD, pacemakers, neurostimulators and other such devices will be excluded.
5. Persons with claustrophobia are excluded.
6. Persons with questionable ferrous implants, bullets, BB's, and shrapnel will be excluded.
7. Subjects who are not fluent in English will be excluded because immediate cooperation and the ability to respond to instructions from the investigators are necessary.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adults with Glut1 Deficiency; Normal, healthy adolescents and adults.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Select metabolite abundance measured at 7Tfield strength | Day 1, immediately after 13 C labeled isotope infusion
  Relative spectral amplitude at equilibrium time point (equilibrium will be defined from the spectra) of the lactate, glucose and bicarbonate spectral peaks arising from infused 13C glucose as measured by magnetic resonance spectroscopy (non contrast brain MRS 7T)
Select metabolite abundance measured at 3T field strength | Day 1, immediately after 13 C labeled isotope infusion
  Relative spectral amplitude at equilibrium time point (equilibrium will be defined from the spectra) of the lactate, glucose and bicarbonate spectral peaks arising from infused 13C glucose as measured by magnetic resonance spectroscopy (non contrast brain MRS 3T)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States